CLINICAL TRIAL: NCT06359977
Title: The Effect of Quantitative Electroencephalography Combined With Ultrasound and Sputum Volume on Predicting Weaning Failure in Neurocritical Patients
Brief Title: The Effect of Quantitative EEG Combined With Ultrasound and Sputum Volume on Predicting Weaning Failure
Status: Not yet recruiting | Type: Observational
Sponsor: Qingdao University (Other)
Responsible Party: Principal Investigator, Bo Yao,phD, The department of critical care medicine, Affiliated hospital of Qingdao university, Qingdao University
Other Study IDs: YB-202442
Record Dates: First submitted 2024-04-02; First posted 2024-04-11 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Weaning Failure
Keywords: Quantitative Electroencephalography; ultrasound

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Neurocritical Patients requiring weaning: The population in this study focused on neurocritical patients with endotracheal intubation. The data of quantitative EEG, beside ultrasound and sputum volume are all recorded for predicting weaning failure.
  Interventions: Other: Quantitative EEG monitoring and beside ultrasound evaluation

INTERVENTIONS:
Other: Quantitative EEG monitoring and beside ultrasound evaluation — After successful spontaneous breathing trial, neurocritical patients undergo at least 2 hours of quantitative EEG monitoring before extubation. Additionally, bedside ultrasound assesses the thickness and variability of the diaphragm, intercostal muscles, rectus abdominis, transversus abdominis, and external oblique muscles. The sputum volume for the 24 hours prior to extubation is also recorded. Reintubation within 48 hours after extubation is defined as weaning failure.

SUMMARY:
Neurocritical patients often face the need for removal of endotracheal tubes. However, despite following the extubation criteria for general critical ill patients, neurocritical patients still exhibit a higher rate of weaning failure, significantly higher than that of general critical ill patients. The extubation criteria for general critical patients emphasize the assessment of lung conditions. However, neurological critical patients often have less severe lung damage, but factors such as consciousness level and coughing ability may significantly influence extubation. Quantitative EEG serves as an objective tool to reflect consciousness level status, while bedside ultrasound can assess respiratory muscle function. Additionally, sputum volume may reflect the condition of lung condition. Therefore, we believe that combination of these three indicators can better predict the success of extubation for neurocritical patients.

ELIGIBILITY:
Inclusion Criteria:

* Neurocritical patients with endotracheal intubation;
* Successful spontaneous Breathing Trial;
* The patients meet extubation criteria evaluated by clinical physician

Exclusion Criteria:

* Patients whose families have opted for cessation of treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population in this study focused on neurocritical patients with endotracheal intubation. The data of quantitative EEG, beside ultrasound and sputum volume are all recorded for predicting weaning failure.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-04-15 (Estimated); Primary Completion 2025-04-15 (Estimated); Study Completion 2025-05-15 (Estimated)

PRIMARY OUTCOMES:
Quantitative EEG indicators | 2 hours before extubation
  These indicators including amplitude EEG and the proportion of α，β，δ，θ wave
Respiratory muscles thickness in centimeter | 2 hours before extubation
  Muscle thickness was evaluated by ultrasound.
Respiratory muscles thickening fraction (%) | 2 hours before extubation
  Muscle thickening fraction was evaluated by ultrasound. It equals (end-inspiratory thickness - end-expiratory thickness)/end-expiratory thickness × 100%.
Sputum volume in milliliter | 24 hours before extubation
  The amount of sputum

CONTACTS AND LOCATIONS:
Overall Officials: bo yao, Dr., Principal Investigator — The Affiliated Hospital of Qingdao University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Welte TM, Gabriel M, Hopfengartner R, Rampp S, Gollwitzer S, Lang JD, Stritzelberger J, Reindl C, Madzar D, Sprugel MI, Huttner HB, Kuramatsu JB, Schwab S, Hamer HM. Quantitative EEG may predict weaning failure in ventilated patients on the neurological intensive care unit. Sci Rep. 2022 May 4;12(1):7293. doi: 10.1038/s41598-022-11196-7. PMID 35508676
- [Result] Bosel J. Who Is Safe to Extubate in the Neuroscience Intensive Care Unit? Semin Respir Crit Care Med. 2017 Dec;38(6):830-839. doi: 10.1055/s-0037-1608773. Epub 2017 Dec 20. PMID 29262440